CLINICAL TRIAL: NCT01188616
Title: Automated Self-management System to Promote Healthy Eating and Activity in Overweight Children
Brief Title: IT-Supported Early Treatment Of Childhood Overweight
Acronym: HEAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: William Adams, MD, Boston Medical Center
Purpose: Treatment
Other Study IDs: H-24963; R21HD050939-01 (NIH)
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Childhood Obesity; Technology Based Obesity Intervention
Keywords: Childhood Obesity; Obesity Intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Telephone Linked Care-HEAT (TLC-HEAT) — A primary care intervention linked with Telephone Linked Care-HEAT (TLC-HEAT), and delivered through an electronic health record (EHR). The HEAT system will guide children in the early stages of overweight toward healthy weight management and assist the child's parent(s) and primary care provider (PCP) to support the child's efforts.

SUMMARY:
The goal of this exploratory/ developmental study is to develop and evaluate an integrated information system, Healthy Eating and Activity Today (HEAT), for promoting self-care in overweight children. HEAT is comprised of two components: 1)Telephone Linked Care-HEAT (TLC-HEAT), a self-care intervention delivered at home through totally automated telephone conversations; and 2) Primary Care-HEAT (PC-HEAT), a primary care intervention linked with TLC-HEAT and delivered through an electronic health record (EHR). The HEAT system will guide children in the early stages of overweight, i.e., children with Body Mass Index (BMI) 0-3 BMI points above the 95th percentile for age and gender, toward healthy weight management and assist the child's parent(s) and primary care provider (PCP) to support the child's efforts.

DETAILED DESCRIPTION:
For this project we will: 1) develop TLC-HEAT for use by children in the earliest stage of overweight and their parents; 2) integrate TLC-HEAT with an electronic health record to provide child- and parent-reported behavior summaries combined with evidence-based decision support to primary care providers (PCPs) at the point-of-care (PC-HEAT); and 3) conduct a pilot study of the combined HEAT system to explore the appropriateness of conducting a larger, randomized clinical trial in the future.

ELIGIBILITY:
Inclusion Criteria:

* Children will be enrolled in the study if they meet a set of eligibility criteria which includes:

  1. 0-3 BMI points above the 95th %ile for age and gender
  2. age 9-12 years old
  3. a PCP at BMC
  4. an English speaking child and parent (based on interviewer assessment).

Exclusion Criteria:

* Children will be considered ineligible for the study if they:

  1. have a health condition for which dietary recommendations in TLC-HEAT would be contraindicated
  2. have cognitive impairment (not in a mainstream academic class in school)
  3. have a terminal illness, current or former diagnosis of an eating disorder, or other diagnosis that the PCP deems should exclude them from participation
  4. plan to move away from the Boston area in less than 12 months
  5. are participating in another clinical weight treatment program.
* Initial screening will be done by research assistants over the phone.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2005-07; Primary Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Adams, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States